CLINICAL TRIAL: NCT04628390
Title: Low Level 810nm Laser Therapy on Controlling Pain During a First Stage of Orthondontic Treatment
Brief Title: Laser Therapy on Controlling Pain During Orthondontic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Universitaria CIEO (Other)
Responsible Party: Principal Investigator, Jaime Enrique Donado Manotas, DDS, Faculty of Endodontic Director, Fundación Universitaria CIEO
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UniCIEO-laser001
Record Dates: First submitted 2020-11-07; First posted 2020-11-13 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Malocclusion
Keywords: Laser; orthodontic; TIP EDGE
MeSH Terms: conditions — Malocclusion | interventions — Lasers; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Sixty patients (60) will be randomized in a 1: 1 ratio, to either of the two arms of this trial.
  Measurements of the primary outcome variable will be done remotely through a virtual pain monitoring questionnaire through a visual analog scale (Baseline, 12 hours, 24 hours, 48 hours, 72 hours)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients participating in the clinical trial, the statistician in charge of the data analysis and the orthodontist will be blinded to the interventions carried out.
  The investigator in charge of applying the intervention will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The low-power therapeutic diode laser will be applied with a wavelength 810nm ± 15nm, output power 0-2 W CW / 0-4.8 W peak power (pulse mode), for a time of 20 seconds per centimeter at lo along the buccal surface of the root of the upper and lower teeth.
  Interventions: Device: Laser
- Placebo (Placebo Comparator): A simulation of the application of therapeutic laser will be carried out as a placebo effect, for a time of 20 seconds per centimeter along the vestibular surface of the root of the upper and lower teeth.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Laser — The laser application will be carried out only once, immediately after the cementation of the orthodontic appliance.
  Other Names: LLLT
  Arms: Experimental
Other: Placebo — Simulation laser application will be carried out only once, immediately after the cementation of the orthodontic appliance.
  Other Names: Simulation laser
  Arms: Placebo

SUMMARY:
To evaluate the effectiveness of pain reduction on a initial orthodontic treatment by using 810nm Diode laser compared to a placebo. Methods: This study will include two parallels groups, 30 adult patients each (mean age 18 - 40) that will be asked to fill a questionnaire related with pain before starting orthodontic treatment with Tip edge technique. Patients from one of the groups will receive laser therapy on both upper and lower maxillary according to the protocol. The patients from the other group will receive a placebo simulating a laser therapy on both maxillary. After the process, both groups will be checked on different times (12hrs-24hrs-48hrs-72hrs after) by filling a questionnaire related with pain each time.

DETAILED DESCRIPTION:
This is a parallel, double-blind, controlled, single-center clinical trial conducted in systemically healthy subjects requiring orthodontic treatment without extractions at the start of treatment in Bogotá, Colombia.

Sixty patients (60) will be randomized in a 1: 1 ratio, to either of the two arms of this trial.

This study will consist of a single visit by the patient, in this visit the assembly and activation of the upper and lower orthodontic appliances will be carried out.

Measurements of the primary outcome variable will be done remotely through a virtual pain monitoring questionnaire through a visual analog scale (Baseline, 12 hours, 24 hours, 48 hours, 72 hours).

After Screening a computer-generated scrambling code will be used for allocation in blocks of 6 to the two treatments.

The identity of included patients will not be provided to the trial team, in order to preserve the blinded aspect of the trial. The identity of the research treatment associated with each randomization number will be hidden from the trial team and patients. The final analysis is scheduled for when 100% of the patients (60 subjects) reach the 72-hour evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed and dated an informed consent form approved by the IRB in accordance with regulatory and institutional guidelines. This form must be obtained before performing any procedure related to the protocol that is not part of the subject's normal regimen.
* No need extractions
* No need Stripping

Exclusion Criteria:

* Periodontal disease
* Pregnant or lactance
* Medicated patients (analgesic, anti-inflammatory drugs, systemic corticosteroids, and calcium channel blockers)
* Cardiac markpaser

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-20 (Estimated); Primary Completion 2021-01-20 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
Measure the "Change in Orthodontic Pain Levels" | Baseline (before treatment), 12 hours (after the start of treatment), 24 hours (after the start of treatment) 48 hours (after the start of treatment) 72 hours(after the start of treatment)
  The evaluation of the difference in pain levels will be determined as a percentage of change and difference in means of pain levels. The difference and the percentage will be calculated by comparing the baseline pain levels observed between the different follow-up times. A rule of three is applied to determine the percentage of change (%) and a subtraction of the pain averages to calculate the difference. Pain analysis will be performed using the visual analog scale (VAS)

SECONDARY OUTCOMES:
Need for analgesic | Baseline (before treatment), 12 hours (after the start of treatment), 24 hours (after the start of treatment) 48 hours (after the start of treatment) 72 hours(after the start of treatment)
  Frequency and Need after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jaime E. Donado, DDS, Principal Investigator — Fundación universitaria CIEO-UniCIEO
Locations (1):
- Fundación universitaria CIEO - UniCIEO, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ordahan B, Karahan AY, Kaydok E. The effect of high-intensity versus low-level laser therapy in the management of plantar fasciitis: a randomized clinical trial. Lasers Med Sci. 2018 Aug;33(6):1363-1369. doi: 10.1007/s10103-018-2497-6. Epub 2018 Apr 7. PMID 29627888
- [Background] Genc G, Kocadereli I, Tasar F, Kilinc K, El S, Sarkarati B. Effect of low-level laser therapy (LLLT) on orthodontic tooth movement. Lasers Med Sci. 2013 Jan;28(1):41-7. doi: 10.1007/s10103-012-1059-6. Epub 2012 Feb 18. PMID 22350425
- [Background] Sommer AP, Schemmer P, Pavlath AE, Forsterling HD, Mester AR, Trelles MA. Quantum biology in low level light therapy: death of a dogma. Ann Transl Med. 2020 Apr;8(7):440. doi: 10.21037/atm.2020.03.159. PMID 32395484
- [Background] Basso FG, Pansani TN, Turrioni AP, Bagnato VS, Hebling J, de Souza Costa CA. In vitro wound healing improvement by low-level laser therapy application in cultured gingival fibroblasts. Int J Dent. 2012;2012:719452. doi: 10.1155/2012/719452. Epub 2012 Jul 15. PMID 22844284
- [Background] Pereira AN, Eduardo Cde P, Matson E, Marques MM. Effect of low-power laser irradiation on cell growth and procollagen synthesis of cultured fibroblasts. Lasers Surg Med. 2002;31(4):263-7. doi: 10.1002/lsm.10107. PMID 12355572
- [Background] Timberlake GT, Enwemeka CS. An inexpensive, automated instrument for laser irradiation of cultured cells. Photomed Laser Surg. 2004 Jun;22(3):233-9. doi: 10.1089/1549541041438614. PMID 15315731
- [Background] Lirani-Galvao AP, Jorgetti V, da Silva OL. Comparative study of how low-level laser therapy and low-intensity pulsed ultrasound affect bone repair in rats. Photomed Laser Surg. 2006 Dec;24(6):735-40. doi: 10.1089/pho.2006.24.735. PMID 17199474
- [Background] Tecco S, D'Attilio M, Tete S, Festa F. Prevalence and type of pain during conventional and self-ligating orthodontic treatment. Eur J Orthod. 2009 Aug;31(4):380-4. doi: 10.1093/ejo/cjp003. Epub 2009 May 22. PMID 19465738
- [Background] Sousa MV, Pinzan A, Consolaro A, Henriques JF, de Freitas MR. Systematic literature review: influence of low-level laser on orthodontic movement and pain control in humans. Photomed Laser Surg. 2014 Nov;32(11):592-9. doi: 10.1089/pho.2014.3789. Epub 2014 Oct 21. PMID 25335088
- [Background] Seifi M, Shafeei HA, Daneshdoost S, Mir M. Effects of two types of low-level laser wave lengths (850 and 630 nm) on the orthodontic tooth movements in rabbits. Lasers Med Sci. 2007 Nov;22(4):261-4. doi: 10.1007/s10103-007-0447-9. Epub 2007 Mar 3. PMID 17334676